CLINICAL TRIAL: NCT01925560
Title: Tolerance and Utilization of Agave Inulin in Healthy Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Urbana-Champaign (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 13359; 13359 (Other Grant/Funding Number: Ingredion Inc.)
Record Dates: First submitted 2013-04-17; First posted 2013-08-19 (Estimated); Last update posted 2014-05-14 (Estimated); Status verified 2014-05

CONDITIONS: Tolerance

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group A- agave inulin or placebo (Experimental): Participant in this group will receive Agave Inulin dose of 5 or 7.5 grams per day or placebo.
  Interventions: Other: Agave Inulin; Other: Placebo
- Group B- agave inulin or placebo (Experimental): Participants in this group will receive Agave Inulin dose of 5 or 7.5 grams per day or placebo
  Interventions: Other: Agave Inulin; Other: Placebo
- Group C-agave inulin or placebo (Experimental): Participants in this group will receive Agave Inulin dose of 5 or 7.5 grams per day or placebo
  Interventions: Other: Agave Inulin; Other: Placebo

INTERVENTIONS:
Other: Agave Inulin — 3x3 Latin square with 3 periods
Other: Placebo — control- 0 (zero) grams/day inulin

SUMMARY:
The objective of this study is to assess the tolerance and utilization of agave inulin. This will be accomplished through analyses of breath and fecal samples to quantify fermentation end-products- hydrogen, carbon dioxide, and methane will be measured in the breath, and short-chain fatty acids, ammonia, phenol, and indole will be measured in feces. Microbial populations will also be measured in fecal samples.

DETAILED DESCRIPTION:
The objective of this study is to assess the tolerance and utilization of agave inulin. This will be accomplished through analyses of breath and fecal samples to quantify fermentation end-products- hydrogen, carbon dioxide, and methane will be measured in the breath, and short-chain fatty acids, ammonia, phenol, and indole will be measured in feces. Microbial populations will also be measured in fecal samples.

ELIGIBILITY:
Inclusion Criteria:

* have body mass index (BMI) between 18.5 and 29.5 kg/m2
* free of metabolic and gastrointestinal diseases

Exclusion Criteria:

* BMI less than 18.5 or greater than 29.5 kg/m2
* presence of metabolic and gastrointestinal diseases
* pregnant or lactating
* taking medications that impact bowel function

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2013-01; Primary Completion 2013-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Breath gas | 21st day of each treatment period
  On the 21st day of each treatment period, participants will come into the laboratory after an overnight (12 hour) fast and begin breath gas testing. The baseline breath gas sample will occur upon arrive. Breath gas collection will utilize the Quintron EasySampler and tubes. Participants will blow into the EasySampler for 1-2 seconds while inserting a tube into a needle holder that allows the collection of the breath gas. After the baseline sample, the participants will consume their respective treatments. Participants then collect subsequent breath gas samples outside of the laboratory every hour for the next 8 hours. All breath gas samples will then be analyzed for CO2, methane, and H2 gases.
Gastrointestinal tolerance | Daily and weekly
  Participants will complete daily and weekly questionnaires to assess tolerance of up to 7.5 g/d agave inulin. Adults completed a weekly survey while meeting with study personnel. They were asked (Yes or No) if they experienced any of the following gastrointestinal symptoms during the past 7 days: nausea, bloating, gastrointestinal rumblings, gas/flatulence, abdominal pain, diarrhea (watery stools). If yes, they rated the intensity of the symptom as no more than usual (0), somewhat more than usual (1), or much more than usual (2). Participants are provided a journal to complete on their own each day, a questionnaire about their stool characteristics. Participants were asked to score the ease of stool passage using the following scale: 1=very easy, 2=easy, 3=neither easy nor difficult, 4=difficult, 5=very difficult.

SECONDARY OUTCOMES:
Fecal fermentation end products | Days 16-20 of each treatment period
  Fecal samples will be collected on days 16-20 of each treatment period. Participants were provided fecal collection materials (fecal hats, coolers, ice packs, and Ziploc bags). Within 15 minutes of defecation, participants will bring their fecal sample to the designated collection site. Fecal samples will then be processed by a team. Fecal specimens will be aliquoted into containers for fermentation end product analysis (short-chain fatty acids, phenols, indoles, ammonia) and dry matter.
Fecal bacteria | Days 16-20 of each treatment period
  Aliquots of fecal samples will be used to quantify bacteria present within fecal samples.
Gastrointestinal Tolerance | Daily during each 21 day treatment period
  Subjective daily gastrointestinal intolerance symptoms for adult human subjects consuming 0, 5.0, or 7.5 grams of agave inulin in a crossover design will be assessed. Gastrointestinal tolerance was scored using the following scale: 1=absent, 2=mild, 3=moderate, 4=severe. All study participants will have booklets with daily tolerance questionnaires in them. The participants will complete the questionnaires on their own each day.
Weekly Gastrointestinal Tolerance Questions | Weekly during each treatment period
  Adults completed a weekly survey while meeting with study personnel. They were asked (Yes or No) if they experienced any of the following gastrointestinal symptoms during the past 7 days: nausea, bloating, gastrointestinal rumblings, gas/flatulence, abdominal pain, diarrhea (watery stools). If yes, they rated the intensity of the symptom as no more than usual (0), somewhat more than usual (1), or much more than usual (2).
Daily Stool Characteristics | Daily during each 21 day treatment period
  Participants are provided a journal to complete on their own each day, a questionnaire about their stool characteristics. Participants were asked to score the ease of stool passage using the following scale: 1=very easy, 2=easy, 3=neither easy nor difficult, 4=difficult, 5=very difficult.
  Stool consistency was scored using the Bristol stool scale: 1=separate hard lumps, like nuts; 2=sausage-shaped but lumpy; 3=like a sausage but with cracks on surface; 4=Like a sausage or snake, smooth and soft; 5=soft blobs with clear-cut edges; 6=fluffy pieces with ragged edges, mushy; 7=watery, no solid pieces, entirely liquid.
Daily food intake journals | Daily during each 21-day treatment period
  Participants were provided a journal to record their daily food and beverage intake. Each week the participants met with a study personnel for 30 minutes to review the journal and turn it in.

CONTACTS AND LOCATIONS:
Overall Officials: Kelly Swanson, PhD, Principal Investigator — UIUC
Locations (1):
- University of Illinois, Urbana, Illinois, United States

REFERENCES:
- [Derived] Kaczmarek JL, Musaad SM, Holscher HD. Time of day and eating behaviors are associated with the composition and function of the human gastrointestinal microbiota. Am J Clin Nutr. 2017 Nov;106(5):1220-1231. doi: 10.3945/ajcn.117.156380. Epub 2017 Sep 27. PMID 28971851
- [Derived] Holscher HD, Bauer LL, Gourineni V, Pelkman CL, Fahey GC Jr, Swanson KS. Agave Inulin Supplementation Affects the Fecal Microbiota of Healthy Adults Participating in a Randomized, Double-Blind, Placebo-Controlled, Crossover Trial. J Nutr. 2015 Sep;145(9):2025-32. doi: 10.3945/jn.115.217331. Epub 2015 Jul 22. PMID 26203099